CLINICAL TRIAL: NCT05939076
Title: First-line Cryoablation for Early Treatment of Persistent Atrial Fibrillation - a Randomized Study Comparing Early Trigger Isolation Using the Cryoballoon Versus Antiarrhythmic Medication
Brief Title: First-line Cryoablation for Early Treatment of Persistent Atrial Fibrillation
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: The Swedish Research Council (Other Government); Erling-Persson Stiftelse (Unknown); Swedish Heart Lung Foundation (Other); Uppsala University (Other)
Responsible Party: Principal Investigator, Carina Blomstrom Lundqvist, MD, PhD, Senior Consultant, Professor, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CryoStopPersAF
Record Dates: First submitted 2023-06-13; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: atrial fibrillation; ablation; first-line; antiarrhythmics; burden; symptoms
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Multicentre, prospective 1:1 randomized open blinded for evaluation of end point (PROBE) controlled parallel-group superiority trial comparing first-line pulmonary vein isolation (PVI) using the cryoballoon (Arctic Front AdvanceR, Medtronic) and first-line antiarrhythmic drug (AAD) therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomised treatment is open but the outcomes are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryoballoon pulmonary vein isolation (Active Comparator): Cryoballoon (Arctic Front AdvanceR, Medtronic) for pulmonary vein isolation
  Interventions: Device: Pulmonary vein isolation
- Antiarrhythmic drug (Active Comparator): Tablet Dronedarone:- 400 mg twice daily or Tablet Flecainide:- (50-)100 (-200) mg twice daily or slow release (100-)200 mg once daily.
  If these drugs fail or give side effects:
  Tablet Propafenone:- 150 mg 3 times daily increasing to 300 mg twice daily, if necessary max 300 mg three times daily. Dose reduction for patients <70 kg bodyweight.
  Tablet Sotalol:- 80 mg twice daily up to 160 mg twice daily. Dose reduction to half dosage if a creatinine clearance is 30-60 ml/min.
  Interventions: Drug: dronedarone - Multaq™ OR flecainide - Tambocor™ OR propafenone - Rytmonorm™ OR sotalol - Sotacor™

INTERVENTIONS:
Device: Pulmonary vein isolation — Arctic Front™ Cryoballoon Advance, Medtronic, for pulmonary vein isolation
  Arms: Cryoballoon pulmonary vein isolation
Drug: dronedarone - Multaq™ OR flecainide - Tambocor™ OR propafenone - Rytmonorm™ OR sotalol - Sotacor™ — Antiarrhythmic drugs
  Arms: Antiarrhythmic drug

SUMMARY:
The goal of this multicentre, prospective, randomized, open, blinded for evaluation of end point (PROBE) controlled parallel-group superiority trial, is to compare the efficacy of antiarrhythmic drug (AAD) therapy and cryoballoon pulmonary vein isolation (PVI) regarding freedom from atrial fibrillation (%) assessed by an implantable cardiac monitor (ICM), ECG tracing or Holter at 12 months in patients with persistent AF. The main question[s] it aims to answer are:

* Will first-line cryoballoon ablation for PVI compared to AAD, result in 25 % higher freedom from atrial tachyarrhythmias lasting > 6 minutes at 12 months (primary outcome) excluding three months initial blanking period, in patients with symptomatic and recurrent persistent AF?
* Will first-line cryoablation for PVI, compared to AAD result in a superior improvement in health related Quality of Life (HRQoL), AF/AT burden, AF/AT progression and reversion, more reverse atrial remodeling, cognitive function, healthcare utilization with associated costs, better safety, at 12-24-36 months as compared with drug use? Participants will be randomized 1:1 to first-line PVI using the cryoballoon or to first-line antiarrhythmic drug therapy and during 3 years follow-up undergo regular;

  * Continuous ECG monitoring for assessment of first AF recurrence and AF burden using an implantable cardiac monitor,
  * Regular echocardiographic exams for reverse atrial remodelling assessment,
  * HRQoL questionnaires
  * Assessment of cognitive function
  * Atrial fibrillation evaluation regarding structured characterisation and AF progression/regression
  * Assessment of Health care use and costs
  * Safety

DETAILED DESCRIPTION:
The primary goal is to evaluate if early pulmonary vein isolation (PVI) performed with the Arctic Front cryoballoon as first-line therapy is superior to antiarrhythmic drugs (AAD) in preventing atrial arrhythmia recurrences in patients with persistent atrial fibrillation (AF).

The main secondary goal is to evaluate the impact of early invasive intervention on health related quality of life (HRQOL) and symptoms, and on safety in comparison to primary AAD therapy, using generic and disease-specific HRQOL questionnaires and also assess Quality Adjusted Life Years (QALYs) score and EHRA classification of symptoms.

The third goal is to assess the impact of an early intervention on cardiovascular health care use and its relation to AF/AT burden and to assess treatment burden and cost-effectiveness compared to AAD.

Study Design: Multicentre, prospective 1:1 randomized open blinded for evaluation of end point (PROBE) controlled parallel-group superiority trial comparing first-line pulmonary vein isolation (PVI) using the cryoballoon (Arctic Front AdvanceR, Medtronic) and first-line antiarrhythmic drug (AAD) therapy. Patients will be randomized 1:1 to first-line PVI using the cryoballoon or to first-line AAD therapy. A 1:1 block randomization immediately after implantation of an implantable cardiac monitor (ICM ) before run-in.

After fulfilling inclusion criteria and no exclusion criteria, an ICM (Reveal Linq™, Medtronic, Inc., Minneapolis, MN) will be injected subcutaneously for continuous rhythm monitoring during a 2 months "run-in" period prior initiation of allocated treatment, and then during 3 years of follow up. A 6 minutes detection cut-off for AF will be used. Patients and physicians will be blinded to the ICM result. Three month blanking period after treatment will not be included in the analysis. SAEs detected via ICM will be managed independently from the blinding of AF. If the ICM has to be explanted the patient should continue in the study with alternative monitoring tool as defined.

The trial will be performed at 4-5 university centres in Sweden, at 1-2 centres in United Kingdom (UK) and at 4-5 centres in Europe, all with experience in Cryoballoon AF ablation. Each centre will register at least 20 -30 patients for a total of 220 patients.

AAD therapy prescribed by the local investigators and collected by the subjects at a pharmacy as in normal clinical practice. They should be initiated with either dronedarone or flecainide as first options. Dronedarone:- 400 mg twice daily or Flecainide:- (50-)100 (-200) mg twice daily or slow release (100-)200 mg once daily. The 3-month "blanking period" will allow for drug titration and optimization. A change to the other of the two first option AADs guided by lack of efficacy defined by AF related symptoms or intolerable side effects. Thereafter, other AADs may be tested in order; propafenone and sotalol as long as the medication changes is within the 3 months blanking period: Propafenone:- 150 mg three times daily increasing to 300 mg twice daily, if necessary max 300 mg three times daily. Sotalol:- 80 mg twice daily up to 160 mg twice daily. Once the blanking period has ended, a change in medication will be defined as clinical endpoint, i.e. treatment failure.

Surveillance of proarrhythmia risk by analysing ECG for prolonged corrected QT interval (QTc), widened QRS-complex, and prolonged PR interval at each follow-up. ECG monitoring on days 1-3 in patients prescribed flecainide, propafenone, or sotalol is recommended. Cardioversion should be performed as soon as possible with adequate protection against thromboembolism if at risk.

Physicians advised to keep patients in the same treatment arm during follow-up. If symptoms worsen despite AAD therapy due to limited efficacy at adequate dosages, the patient may, if requested, undergo AF ablation with PVI following preferably a minimum of 12 months AAD therapy.

Catheter ablation with PVI should follow clinical routine. PVI alone will be performed using a 28 mm cryoballoon with an Achieve circular mapping (ACM) catheter for recording of pulmonary vein potentials. Cryoballoon application for 4 minutes in each vein guided by disappearance of PV potentials or by reduction of temperature to at least minus 40 C degrees within the first 120 seconds if no PV potentials can be visualized. After ablation of all pulmonary veins, entrance block during sinus rhythm should be assessed with PV entrance block documented from each PV using a circular mapping catheter.

Biomarkers s100b, troponin-T (TnT) and NT-pro-BNP (brain natriuretic peptide) will be obtained from peripheral venous blood in the lab on the day of the procedure (baseline) before placing the catheters in the heart and again after all ablation applications after the transseptal catheter has been withdrawn. All three markers are thereafter sampled a third time from peripheral blood after 6-18 hours, and NT-pro-BNP at 3, 12, 24, 36 months follow up.

Follow-up Re-ablations may be performed at earliest 3 months after the prior AF ablation procedure if symptoms persists or recurs provided an AF/AT is ECG documented. PVI alone will be performed using a cryoballoon with a circular mapping catheter for assessing entrance conduction block. Patients may be offered a 3rd AF ablation. If patient declines a repeat intervention despite symptomatic recurrence of AF, the patient may be offered AAD, and will be defined as failed ablation unless a beta-blocking agent alone is prescribed. If all PVs are isolated at a repeat ablation procedure, other lesions may be performed except for posterior wall isolation unless pulsed field ablation is used, but treatment will be defined as failed PVI.

The study duration is 3 years with 18 months' enrolment period. Patients will be followed at three, six, nine, 12, 18, 24, 30 and 36 months after the ablation procedure or start of AAD therapy. A nurse telephone visit will be scheduled at 6, 9, 18 and 30 months for recording of clinical events, medication and adverse events. All endpoints will be evaluated at last visit before cross-over.

A clinical event is any event related to a cardiovascular disease or AF/AT; such as acquisition of a new comorbidity, new risk factor that results in increased bleeding risk, new cardiovascular intervention such as cardioversion, angiography, bypass surgery etc but which is not defined as an AE.

All "Serious Adverse Events" (SAE) will be documented on the "Adverse events Form" AND "Serious adverse events Form" and reported to an independent Clinical Events Committee. All deaths events will be documented on "Death report forms".All-cause death will be classified as either Non-cardiovascular (including unknown, excluding sudden death or Cardiovascular death (Cardiac (sudden (including arrhythmic, myocardial infarction) vs non-sudden) or Vascular) Statistical analysis Safety - All randomized patients will be included in the safety analysis. Only observed observations are used in the safety analysis.

Modified Intention to treat (mITT) - All randomized patients who receive treatment. The main analysis will be performed on the mITT-population.

Per protocol (PP) - All randomized patients completing the study treatment period of 12 months without any major protocol violation (for example ineligibility, early withdrawals, poor compliance). The PP population will be defined at clean file.

Missing Data; The Primary variable will be imputed using a "worst case imputation" for the Logistic Regression if the magnitude of the missing data is small, say, approximately 5%. The Statistical Analysis Plan will include an outline for the multiple imputation strategy to be used for the situation with a larger amount of missing primary endpoints.

The hypothesis generating analyses of Secondary Variables will use a simplistic Last Observation approach in case the amount of missing data is limited, say, less than 5%. The Statistical analysis Plan (SAP) will include an outline for the multiple imputation strategy to be used for the situation with a larger amount of missing secondary endpoints.

Subgroups and explorative analyses; Explorative analyses may be performed to investigate relationships between treatments and endpoints, and for predictive factors for AF recurrences.

Statistical methods; The Primary variable, freedom from atrial tachyarrhythmia at least 12 months with 90-day initial blanking period, will be analyzed using a Logistic Regression adjusted for the following additional covariates (baseline values): Coronary artery disease, Hypertension and left atrial volume index. Graphical methods such as Kaplan-Meier plots will be used to visualize the treatment effect in the full study population: "Freedom of tachyarrhythmia up to 12 months with 90-day blanking period".

The main analysis population will be a modified Intention to Treat population: all treated patients as randomized. The number of randomized subjects who are not treated are assumed to be at most a handful. The Per Protocol population will be defined at the Clean File Meeting and will be used for sensitivity analysis for the analysis of the primary variable using the same methods as for the main analysis.

The set of secondary variables will not be adjusted for multiplicity. All findings among secondary variables in main population viewed as exploratory and hypothesis generating. The statistical Methods for each of the Secondary Endpoints will be described in detail in the Statistical Analysis Plan. All continuous variables will be presented per treatment group using descriptive statistics by mean, standard deviation (SD), max and min values, in addition medians, 25th and 75th percentiles will be presented when suitable. The mean difference between treatment groups will be presented with 95% Confidence Intervals (CIs).

Sample Calculation: Study randomized 1:1: Proportion of freedom from atrial tachy-arrhythmia before 12 months with 90-day blanking period estimated to reach 55% in Ablation group based on previous cryoballoon AF ablation study of persistent AF patients monitored by ICM versus 30% in Drug arm, based on 25% difference in freedom from AF between treatment groups in a first line treatment study of paroxysmal AF patients. The 40% freedom from AF postablation in persist AF patients judged too pessimistic for a first line trial. Three prior AAD trials evaluating drug efficacy in persistent AF patients post cardioversion, using intermittent recordings, reported freedom from AF ranging between 30 and 42 %. Recognising that ICM would detect more AF episodes, the freedom from AF post cardioversion on AAD at 12 months is therefore estimated to be in the lower range, i.e. 30 %, in this trial.

A 2 minutes AF detection cut-off has a lower positive predictive value versus a 6 min cut-off episode duration, which will decrease number of total episode count and false positive detection without neglecting relevant clinical information, keeping AF-burden unaffected. It therefore seems rational to use 6 minutes as AF episode cut-off, which is anticipated to at most increase the freedom from AF by 5% in both treatment groups but without affecting the relative treatment differences in the 2 groups.

To have a 90% chance (i.e. power=90%) at the 5% significance level of detecting an improvement in the primary outcome from 30% in the control group to 55% in the ablation group, a total of 156 patients are needed. Adjusting for an assumed cross over rate of approximately 10% in the drug arm and 5% in the Ablation arm the total sample size will be 220.

Treatment allocation sequence generated in Statistical Analysis Software (SAS) or R by the Biostatistics section at Uppsala Clinical Research Centre (UCR) by using permuted blocks and 1:1 allocation, stratification by center and type of persistent AF. Patients randomized using the Interactive Web Response System (IWRS) function in Viedoc.

ELIGIBILITY:
Inclusion Criteria:

* Non-longstanding persistent symptomatic AF with at least 2 episodes within last 24 months, the latest episode within the previous 6 months and one documented on a 12 lead ECG or Holter monitor, that is classified as either

  1. Classical persistent AF (continuously sustained beyond 7 days and <12 months in duration) as defined by ESC guidelines14 OR
  2. Persistent AF which has progressed from paroxysmal AF (patients who have been cardioverted within 7 days of onset provided a history of spontaneous conversion to sinus rhythm is lacking during the past 24 months).
* Candidate for rhythm control therapy; AF ablation or AAD based on symptomatic AF.

Exclusion Criteria:

1. Regular daily use of AAD class I or III at adequate therapeutic dosages (pill-in-the-pocket permitted, beta-blockers permitted).
2. Previous AF ablation or surgery.
3. Severe heart failure (NYHA III-IV).
4. Reduced left ventricular ejection fraction (LVEF ≤40 % during sinus rhythm).
5. Hypertrophic cardiomyopathy (septal or posterior wall thickness >1.5 cm)
6. Severely enlarged LA with left atrial volume indexed to body surface area (LAVI, ml/m2) > 48.
7. Significant valvular disease requiring treatment or valve prothesis.
8. Severe Chronic Obstructive Pulmonary Disease (COPD) stage III or chronic kidney disease (eGFR< 30 umol/l)).
9. Planned cardiac intervention within the next 12 months or cardiac surgery last 6 months.
10. Myocardial infarction, revascularisation previous 6 months.
11. Stroke or Transient Ischemic Attack (TIA) within previous 6 months.
12. Tachycardiomyopathy.
13. Dependent on VVI (ventricular single chamber inhibited) pacing.
14. Conventional contraindications for AF ablation including AF due to reversible causes and contraindications for both class IC and class III antiarrhythmic drugs.
15. Expected survival less than 3 years, alcohol or drug abuse.
16. Participation in another trial or absence of consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-08-21 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients free from first atrial tachyarrhythmia recurrence lasting 6 minutes or longer | 12 months after initiation of allocated treatment excluding the first 3 months blanking period
  In the absence of antiarrhythmic drugs in ablation group as documented by an implantable cardiac monitor from initiation of treatment.

SECONDARY OUTCOMES:
Total atrial arrhythmia burden (percentage of time in AF/AT) | baseline,12, 24, 36 months after initiation of treatment excluding the 3 months blanking period
  Measured from the continuous implantable cardiac monitor with a 6 minutes AF episode detection cut-off limit.
AF progression and reversion | baseline,12, 24, 36 months follow-up excluding 3 months blanking period
  Progression to longstanding persistent or permanent AF/AT and regression going in opposite direction from persistent to paroxysmal AF or to sinus rhythm. Measured as combination of reduced number of progressions or increased number of AF/AT regression .
Generic Health Related Quality of life (HRQoL) | baseline, 12, 24, 36 months follow-up
  Generic Medical Outcomes Study Short Form-36 (SF-36) quality of life questionnaire using 8 subscales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Scores from 0 to 100; lower scores poorer QoL.
Symptoms | baseline, 12, 24, 36 months after initiation of treatment
  European Heart Rhythm Association (EHRA) Symptom Classification assessing the severity of AF related symptoms
AF specific Health Related Quality of Life | baseline, 12, 24, 36 months after initiation of treatment excluding the 3 months blanking period
  Assessed by University of Toronto Atrial Fibrillation Severity Scale (AFSS); 19-item AF-specific scale; ratings AF including 4 categories;
  1. AF burden (calculated from modified sum of frequency, duration and severity of episodes); Total AF Burden=AF frequency + AF duration + AF severity. Each of 3 measures contributes equally to Total AF Burden score, and varies from 1-10 to yield Total AF Burden scores ranging from 3-30 where higher scores indicate greater AF burden.
  2. Global Well Being (visual analogue scale 1-10; worst - best possible life);
  3. AF Symptom Score (sum of 7 items on specified symptoms); For each of 7 questions (answers vary from 0=I have not had this symptom in past 4 weeks to 5=A great deal), values determined and summed together to form a total score (0-35). This score assumes linearity of severity.
  4. Health Care Utilization (number of cardioversions, ablations, emergency room visits, hospitalizations due to arrhythmia, and specialist appointments).
Cognitive function | baseline,12, 24, 36 months after initiation of treatment
  Trail Making Test (TMT) parts A and B. Patient is asked to draw lines from figures in consecutive orders n 1-2-3 etc (TMT A) and from figures to letters 1-A-2-B etc.(TMT B) Examiner starts timing both part A and B and counts errors made. The Time in seconds and Number of errors are counted for both A and B test. The rhythm and pulse at the time of the evaluation will be recorded but is not used as a measure other than a binary value for correlation with cognitive function.
Rate of Healthcare utilizations for cardiovascular reasons | baseline,12, 24, 36 months after initiation of treatment excluding the 3 months blanking period
  Number of cardioversions, ablations, drug initiations, cardiovascular hospitalizations, emergency department visits and unplanned outpatient visits and its relation to AF/AT burden.
  Cardiovascular means related to AF including any treatment or diagnostic procedure for AF/AT, i.e. cardioversions, medication, further AF ablations after AF/AT recurrence, or any adverse events related to AF/AT or its treatment (acute stroke), heart failure, myocardial ischemic events; adverse events (eg. pacemaker implantation).
Cost-effectiveness analysis by EuroQol-5 Dimensions (EQ-5D) | 36 months
  Quality-adjusted life years (QALYs) using EQ-5D; QALYs will then be incorporated with medical costs; cost/QALY to compare the treatments.
  i) EQ-5D descriptive system with five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, each with 5 levels. Digits combined into a 5-digit number for patient's health state.
  ii) Visual analogue vertical line scale (EQ-VAS) with endpoints labelled 'The best and worst health you can imagine' as a quantitative measure of health outcome reflecting patient's own judgement.
  Cost-effectiveness analysis of the treatments examining costs and health outcomes of the two interventions. It compares the interventions by estimating how much it costs to gain a unit of a health outcome.
Proportion of patients with Reverse atrial remodeling | baseline, 12, 24 and 36 months
  Proportion of patients with Reverse atrial remodeling as defined by at least 15% decrease of Left atrial maximal volume index (ml/m2) or increase of left atrial strain during reservoir phase (percentage) or left atrial strain during contraction phase (percentage) versus baseline.
Proportion of patients free from ECG documented atrial tachyarrhythmia recurrence lasting 6 minutes or longer after the 1st and last ablation procedure respectively | 36 months
  Defined as single and multiple procedure success
Adverse events | 12, 24, 36 months
  Type and frequency of adverse events and serious adverse events related or not to treatment.
Numbers of withdrawals / 'cross-overs' | 12, 24, 36 months
  Frequency of withdrawals / 'cross-overs' in each treatment group
Covariate adjusted primary endpoint freedom from first atrial tachyarrhythmia recurrence lasting 6 minutes or longer | 12 and 36 months
  Analysis using following covariates at baseline: coronary artery disease, hypertension, left atrial volume index.

OTHER OUTCOMES:
Predictors of non-responders by 4-Structured - AF characterization and conventional risk factors | 12 and 24 months
  Structured AF (4S-AF) characterization assessing;
  1. Stroke risk; No Oral Anticoagulation (OAC) or OAC = 0 - 1 point.
  2. Symptom severity by European Heart Rhythm Association (EHRA) Symptom (0 point = EHRA score 1-2a; 1 point = EHRA score 2b; 2 points = EHRA score 3-4).
  3. Severity AF/AT burden (0 point = short, infrequent, 1 point = intermediate and/or frequent; 2 points = long or very frequent).
  4. Substrate: Comorbidity/Left atrial enlargement (0 point = none; 1 = single/mild moderate; 2 points = multiple/ severe). Add +1 point if age >75 years.
  Sum of points will be correlated to treatment responder, defined as sinus rhythm at 12 months without AF/AT recurrences, versus conventional.
  Conventional risk factors for AF/AT recurrence:
  1. AF history, (months)
  2. P wave duration (milliseconds)
  3. LAVI (mL/m2) and atrial strain (percentage) by echocardiography
  4. NTpro-BNP (ng/L)
  5. BMI (kg/m2)
  6. CHA2DS2vasc score (0-10)
Blood pressure, systolic | baseline,12, 24, 36 months after initiation of treatment
  Measured after 10 minutes rest by (mmHg).
Blood pressure, diastolic (mmHg). | baseline,12, 24, 36 months after initiation of treatment
  Measured after 10 minutes rest by (mmHg).
Rhythm at time of responding to quality of life questionnaire | baseline, 12, 24, 36 months
  Rhythm (atrial fibrillation or sinus rhythm) recorded at time of quality of life assessment for evaluation if correlated to QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Carina M Blomstrom Lundqvist, MD, PhD, Principal Investigator — Faculty of Medicine and Health, Örebro University, and Uppsala University, Sweden
Locations (6):
- Electrophysiology Department, Heart Institute, University of Pecs, Pécs, Hungary
- Div. of Arrhythmia and Pacing, National Cardiovascular Institute, Faculty of Medicine, Slovak Medical University, Bratislava, Slovakia
- Sweden (3):
  - Institute of Medicine. Sahlgrenska Academy at University of Gothenburg, Gothenburg
  - Department of Cardiology, School of Medical Sciences, Faculty of Medicine and Health, Örebro University, Örebro
  - Department of Medical Science, Uppsala University Hospital, Uppsala
- Department of Cardiac Electrophysiology, Liverpool Centre for Cardiovascular Science, University of Liverpool and Liverpool Heart & Chest Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Restrictions related to Review Ethical Boards

REFERENCES:
- [Background] Wazni OM, Dandamudi G, Sood N, Hoyt R, Tyler J, Durrani S, Niebauer M, Makati K, Halperin B, Gauri A, Morales G, Shao M, Cerkvenik J, Kaplon RE, Nissen SE; STOP AF First Trial Investigators. Cryoballoon Ablation as Initial Therapy for Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):316-324. doi: 10.1056/NEJMoa2029554. Epub 2020 Nov 16. PMID 33197158
- [Background] Kuniss M, Pavlovic N, Velagic V, Hermida JS, Healey S, Arena G, Badenco N, Meyer C, Chen J, Iacopino S, Anselme F, Packer DL, Pitschner HF, Asmundis C, Willems S, Di Piazza F, Becker D, Chierchia GB; Cryo-FIRST Investigators. Cryoballoon ablation vs. antiarrhythmic drugs: first-line therapy for patients with paroxysmal atrial fibrillation. Europace. 2021 Jul 18;23(7):1033-1041. doi: 10.1093/europace/euab029. PMID 33728429
- [Background] Wazni OM, Marrouche NF, Martin DO, Verma A, Bhargava M, Saliba W, Bash D, Schweikert R, Brachmann J, Gunther J, Gutleben K, Pisano E, Potenza D, Fanelli R, Raviele A, Themistoclakis S, Rossillo A, Bonso A, Natale A. Radiofrequency ablation vs antiarrhythmic drugs as first-line treatment of symptomatic atrial fibrillation: a randomized trial. JAMA. 2005 Jun 1;293(21):2634-40. doi: 10.1001/jama.293.21.2634. PMID 15928285
- [Background] Morillo CA, Verma A, Connolly SJ, Kuck KH, Nair GM, Champagne J, Sterns LD, Beresh H, Healey JS, Natale A; RAAFT-2 Investigators. Radiofrequency ablation vs antiarrhythmic drugs as first-line treatment of paroxysmal atrial fibrillation (RAAFT-2): a randomized trial. JAMA. 2014 Feb 19;311(7):692-700. doi: 10.1001/jama.2014.467. PMID 24549549
- [Background] Cosedis Nielsen J, Johannessen A, Raatikainen P, Hindricks G, Walfridsson H, Kongstad O, Pehrson S, Englund A, Hartikainen J, Mortensen LS, Hansen PS. Radiofrequency ablation as initial therapy in paroxysmal atrial fibrillation. N Engl J Med. 2012 Oct 25;367(17):1587-95. doi: 10.1056/NEJMoa1113566. PMID 23094720
- [Background] De Greef Y, Schwagten B, Chierchia GB, de Asmundis C, Stockman D, Buysschaert I. Diagnosis-to-ablation time as a predictor of success: early choice for pulmonary vein isolation and long-term outcome in atrial fibrillation: results from the Middelheim-PVI Registry. Europace. 2018 Apr 1;20(4):589-595. doi: 10.1093/europace/euw426. PMID 28340103
- [Background] Kawaji T, Shizuta S, Yamagami S, Aizawa T, Komasa A, Yoshizawa T, Kato M, Yokomatsu T, Miki S, Ono K, Kimura T. Early choice for catheter ablation reduced readmission in management of atrial fibrillation: Impact of diagnosis-to-ablation time. Int J Cardiol. 2019 Sep 15;291:69-76. doi: 10.1016/j.ijcard.2019.03.036. Epub 2019 Mar 20. PMID 30948218
- [Background] Hussein AA, Saliba WI, Barakat A, Bassiouny M, Chamsi-Pasha M, Al-Bawardy R, Hakim A, Tarakji K, Baranowski B, Cantillon D, Dresing T, Tchou P, Martin DO, Varma N, Bhargava M, Callahan T, Niebauer M, Kanj M, Chung M, Natale A, Lindsay BD, Wazni OM. Radiofrequency Ablation of Persistent Atrial Fibrillation: Diagnosis-to-Ablation Time, Markers of Pathways of Atrial Remodeling, and Outcomes. Circ Arrhythm Electrophysiol. 2016 Jan;9(1):e003669. doi: 10.1161/CIRCEP.115.003669. PMID 26763227
- [Background] Irfan G, de Asmundis C, Mugnai G, Poelaert J, Verborgh C, Umbrain V, Beckers S, Hacioglu E, Hunuk B, Velagic V, Stroker E, Brugada P, Chierchia GB. One-year follow-up after second-generation cryoballoon ablation for atrial fibrillation in a large cohort of patients: a single-centre experience. Europace. 2016 Jul;18(7):987-93. doi: 10.1093/europace/euv365. Epub 2015 Dec 23. PMID 26705562
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Gallagher C, Hendriks JM, Giles L, Karnon J, Pham C, Elliott AD, Middeldorp ME, Mahajan R, Lau DH, Sanders P, Wong CX. Increasing trends in hospitalisations due to atrial fibrillation in Australia from 1993 to 2013. Heart. 2019 Sep;105(17):1358-1363. doi: 10.1136/heartjnl-2018-314471. Epub 2019 Apr 1. PMID 30936408
- [Background] Andrade J, Khairy P, Dobrev D, Nattel S. The clinical profile and pathophysiology of atrial fibrillation: relationships among clinical features, epidemiology, and mechanisms. Circ Res. 2014 Apr 25;114(9):1453-68. doi: 10.1161/CIRCRESAHA.114.303211. PMID 24763464
- [Background] Singh BN, Singh SN, Reda DJ, Tang XC, Lopez B, Harris CL, Fletcher RD, Sharma SC, Atwood JE, Jacobson AK, Lewis HD Jr, Raisch DW, Ezekowitz MD; Sotalol Amiodarone Atrial Fibrillation Efficacy Trial (SAFE-T) Investigators. Amiodarone versus sotalol for atrial fibrillation. N Engl J Med. 2005 May 5;352(18):1861-72. doi: 10.1056/NEJMoa041705. PMID 15872201
- [Background] Chun KJ, Byeon K, Im SI, Park KM, Park SJ, Kim JS, On YK. Efficacy of dronedarone versus propafenone in the maintenance of sinus rhythm in patients with atrial fibrillation after electrical cardioversion. Clin Ther. 2014 Sep 1;36(9):1169-75. doi: 10.1016/j.clinthera.2014.07.013. Epub 2014 Aug 16. PMID 25134972
- [Background] Alegret JM, Vinolas X, Grande A, Castellanos E, Asso A, Tercedor L, Carmona JR, Medina O, Alberola AG, Fidalgo ML, Perez-Alvarez L, Sabate X. Clinical effectiveness of antiarrhythmic treatment after electrical cardioversion in patients without structural heart disease. Rev Esp Cardiol. 2008 Dec;61(12):1274-9. doi: 10.1016/s1885-5857(09)60055-4. English, Spanish. PMID 19080966
- [Background] Le Heuzey JY, De Ferrari GM, Radzik D, Santini M, Zhu J, Davy JM. A short-term, randomized, double-blind, parallel-group study to evaluate the efficacy and safety of dronedarone versus amiodarone in patients with persistent atrial fibrillation: the DIONYSOS study. J Cardiovasc Electrophysiol. 2010 Jun 1;21(6):597-605. doi: 10.1111/j.1540-8167.2010.01764.x. Epub 2010 Apr 6. PMID 20384650
- [Background] Gwag HB, Chun KJ, Hwang JK, Park SJ, Kim JS, Park KM, On YK. Which antiarrhythmic drug to choose after electrical cardioversion: A study on non-valvular atrial fibrillation patients. PLoS One. 2018 May 22;13(5):e0197352. doi: 10.1371/journal.pone.0197352. eCollection 2018. PMID 29787592
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Malmborg H, Lonnerholm S, Blomstrom P, Blomstrom-Lundqvist C. Ablation of atrial fibrillation with cryoballoon or duty-cycled radiofrequency pulmonary vein ablation catheter: a randomized controlled study comparing the clinical outcome and safety; the AF-COR study. Europace. 2013 Nov;15(11):1567-73. doi: 10.1093/europace/eut104. Epub 2013 May 22. PMID 23703361
- [Background] Blomstrom-Lundqvist C, Gizurarson S, Schwieler J, Jensen SM, Bergfeldt L, Kenneback G, Rubulis A, Malmborg H, Raatikainen P, Lonnerholm S, Hoglund N, Mortsell D. Effect of Catheter Ablation vs Antiarrhythmic Medication on Quality of Life in Patients With Atrial Fibrillation: The CAPTAF Randomized Clinical Trial. JAMA. 2019 Mar 19;321(11):1059-1068. doi: 10.1001/jama.2019.0335. PMID 30874754
- [Background] Packer DL, Mark DB, Robb RA, Monahan KH, Bahnson TD, Poole JE, Noseworthy PA, Rosenberg YD, Jeffries N, Mitchell LB, Flaker GC, Pokushalov E, Romanov A, Bunch TJ, Noelker G, Ardashev A, Revishvili A, Wilber DJ, Cappato R, Kuck KH, Hindricks G, Davies DW, Kowey PR, Naccarelli GV, Reiffel JA, Piccini JP, Silverstein AP, Al-Khalidi HR, Lee KL; CABANA Investigators. Effect of Catheter Ablation vs Antiarrhythmic Drug Therapy on Mortality, Stroke, Bleeding, and Cardiac Arrest Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1261-1274. doi: 10.1001/jama.2019.0693. PMID 30874766
- [Background] Mortsell D, Jansson V, Malmborg H, Lonnerholm S, Blomstrom-Lundqvist C. Clinical outcome of the 2nd generation cryoballoon for pulmonary vein isolation in patients with persistent atrial fibrillation - A sub-study of the randomized trial evaluating single versus dual cryoballoon applications. Int J Cardiol. 2019 Mar 1;278:120-125. doi: 10.1016/j.ijcard.2018.10.097. Epub 2018 Oct 29. PMID 30409738
- [Background] Tilz RR, Rillig A, Thum AM, Arya A, Wohlmuth P, Metzner A, Mathew S, Yoshiga Y, Wissner E, Kuck KH, Ouyang F. Catheter ablation of long-standing persistent atrial fibrillation: 5-year outcomes of the Hamburg Sequential Ablation Strategy. J Am Coll Cardiol. 2012 Nov 6;60(19):1921-9. doi: 10.1016/j.jacc.2012.04.060. Epub 2012 Oct 10. PMID 23062545
- [Background] B Schnabel R, Pecen L, Engler D, Lucerna M, Sellal JM, Ojeda FM, De Caterina R, Kirchhof P. Atrial fibrillation patterns are associated with arrhythmia progression and clinical outcomes. Heart. 2018 Oct;104(19):1608-1614. doi: 10.1136/heartjnl-2017-312569. Epub 2018 Mar 17. PMID 29550771
- [Background] de Vos CB, Pisters R, Nieuwlaat R, Prins MH, Tieleman RG, Coelen RJ, van den Heijkant AC, Allessie MA, Crijns HJ. Progression from paroxysmal to persistent atrial fibrillation clinical correlates and prognosis. J Am Coll Cardiol. 2010 Feb 23;55(8):725-31. doi: 10.1016/j.jacc.2009.11.040. PMID 20170808
- [Background] Ogawa H, An Y, Ikeda S, Aono Y, Doi K, Ishii M, Iguchi M, Masunaga N, Esato M, Tsuji H, Wada H, Hasegawa K, Abe M, Lip GYH, Akao M; Fushimi AF Registry Investigators. Progression From Paroxysmal to Sustained Atrial Fibrillation Is Associated With Increased Adverse Events. Stroke. 2018 Oct;49(10):2301-2308. doi: 10.1161/STROKEAHA.118.021396. PMID 30355097
- [Background] J Albano A, Bush J, L Parker J, Corner K, W Lim H, P Brunner M, I Dahu M, Dandamudi S, Elmouchi D, Gauri A, Woelfel A, Chalfoun NT. Left Atrial Volume Index Predicts Arrhythmia-Free Survival in Patients with Persistent Atrial Fibrillation Undergoing Cryoballoon Ablation. J Atr Fibrillation. 2019 Aug 31;12(2):2192. doi: 10.4022/jafib.2192. eCollection 2019 Aug-Sep. PMID 32002112
- [Background] Csecs I, Yamaguchi T, Kheirkhahan M, Czimbalmos C, Fochler F, Kholmovski EG, Morris AK, Kaur G, Vago H, Merkely B, Chelu MG, Marrouche NF, Wilson BD. Left atrial functional and structural changes associated with ablation of atrial fibrillation - Cardiac magnetic resonance study. Int J Cardiol. 2020 Apr 15;305:154-160. doi: 10.1016/j.ijcard.2019.12.010. Epub 2019 Dec 6. PMID 31874788
- [Background] Costa FM, Ferreira AM, Oliveira S, Santos PG, Durazzo A, Carmo P, Santos KR, Cavaco D, Parreira L, Morgado F, Adragao P. Left atrial volume is more important than the type of atrial fibrillation in predicting the long-term success of catheter ablation. Int J Cardiol. 2015 Apr 1;184:56-61. doi: 10.1016/j.ijcard.2015.01.060. Epub 2015 Jan 27. PMID 25697871
- [Background] Walters TE, Nisbet A, Morris GM, Tan G, Mearns M, Teo E, Lewis N, Ng A, Gould P, Lee G, Joseph S, Morton JB, Zentner D, Sanders P, Kistler PM, Kalman JM. Progression of atrial remodeling in patients with high-burden atrial fibrillation: Implications for early ablative intervention. Heart Rhythm. 2016 Feb;13(2):331-9. doi: 10.1016/j.hrthm.2015.10.028. Epub 2015 Oct 17. PMID 26484789
- [Background] Scherschel K, Hedenus K, Jungen C, Lemoine MD, Rubsamen N, Veldkamp MW, Klatt N, Lindner D, Westermann D, Casini S, Kuklik P, Eickholt C, Klocker N, Shivkumar K, Christ T, Zeller T, Willems S, Meyer C. Cardiac glial cells release neurotrophic S100B upon catheter-based treatment of atrial fibrillation. Sci Transl Med. 2019 May 22;11(493):eaav7770. doi: 10.1126/scitranslmed.aav7770. PMID 31118294
- [Background] Antman EM, Tanasijevic MJ, Thompson B, Schactman M, McCabe CH, Cannon CP, Fischer GA, Fung AY, Thompson C, Wybenga D, Braunwald E. Cardiac-specific troponin I levels to predict the risk of mortality in patients with acute coronary syndromes. N Engl J Med. 1996 Oct 31;335(18):1342-9. doi: 10.1056/NEJM199610313351802. PMID 8857017
- [Background] Sawhney V, Schilling RJ, Providencia R, Cadd M, Perera D, Chatha S, Mercer B, Finlay M, Halimi F, Pavin D, Anselme F, Cebron JP, Chun J, Schmidt B, Defaye P, Dhillon G, Boveda S, Albenque JP, Tayebjee M, de Asmundis C, Chierchia G, Hunter RJ. Cryoablation for persistent and longstanding persistent atrial fibrillation: results from a multicentre European registry. Europace. 2020 Mar 1;22(3):375-381. doi: 10.1093/europace/euz313. PMID 31808520
- [Background] Chun KR, Stich M, Furnkranz A, Bordignon S, Perrotta L, Dugo D, Bologna F, Schmidt B. Individualized cryoballoon energy pulmonary vein isolation guided by real-time pulmonary vein recordings, the randomized ICE-T trial. Heart Rhythm. 2017 Apr;14(4):495-500. doi: 10.1016/j.hrthm.2016.12.014. Epub 2016 Dec 9. PMID 27956248
- [Background] Bollmann A, Ueberham L, Schuler E, Wiedemann M, Reithmann C, Sause A, Tebbenjohanns J, Schade A, Shin DI, Staudt A, Zacharzowsky U, Ulbrich M, Wetzel U, Neuser H, Bode K, Kuhlen R, Hindricks G. Cardiac tamponade in catheter ablation of atrial fibrillation: German-wide analysis of 21 141 procedures in the Helios atrial fibrillation ablation registry (SAFER). Europace. 2018 Dec 1;20(12):1944-1951. doi: 10.1093/europace/euy131. PMID 29982554
- [Background] Oikawa J, Fukaya H, Wada T, Horiguchi A, Kishihara J, Satoh A, Saito D, Sato T, Matsuura G, Arakawa Y, Kobayashi S, Shirakawa Y, Nishinarita R, Ishizue N, Katada C, Tanabe S, Niwano S, Ako J. Additional posterior wall isolation is associated with gastric hypomotility in catheter ablation of atrial fibrillation. Int J Cardiol. 2021 Mar 1;326:103-108. doi: 10.1016/j.ijcard.2020.10.069. Epub 2020 Oct 31. PMID 33130261
- [Background] Sulke N, Dulai R, Freemantle N, Sugihara C, Podd S, Eysenck W, Lewis M, Hyde J, Veasey RA, Furniss SS. Long Term outcomes of percutaneous atrial fibrillation ablation in patients with continuous monitoring. Pacing Clin Electrophysiol. 2021 Jul;44(7):1176-1184. doi: 10.1111/pace.14282. Epub 2021 Jun 11. PMID 34028066
- [Background] Wechselberger S, Kronborg M, Huo Y, Piorkowski J, Neudeck S, Passler E, El-Armouche A, Richter U, Mayer J, Ulbrich S, Pu L, Kirstein B, Gaspar T, Piorkowski C. Continuous monitoring after atrial fibrillation ablation: the LINQ AF study. Europace. 2018 Nov 1;20(FI_3):f312-f320. doi: 10.1093/europace/euy038. PMID 29688326
- [Result] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916
- [Result] Andrade JG, Wells GA, Deyell MW, Bennett M, Essebag V, Champagne J, Roux JF, Yung D, Skanes A, Khaykin Y, Morillo C, Jolly U, Novak P, Lockwood E, Amit G, Angaran P, Sapp J, Wardell S, Lauck S, Macle L, Verma A; EARLY-AF Investigators. Cryoablation or Drug Therapy for Initial Treatment of Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):305-315. doi: 10.1056/NEJMoa2029980. Epub 2020 Nov 16. PMID 33197159

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT05939076/Prot_SAP_000.pdf